CLINICAL TRIAL: NCT04154423
Title: Comparing Approaches to Enhanced Prenatal Care to Improve Maternal and Child Health in Central CA
Brief Title: Engaging Mothers & Babies; Reimagining Antenatal Care for Everyone (EMBRACE) Study
Acronym: EMBRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); California State University, Fresno Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AD-2018C2-13227
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Premature Birth; Pregnancy Preterm; Prenatal Stress; Depression, Anxiety; Depression, Postpartum; Satisfaction, Patient; Health Problems in Pregnancy
Keywords: Premature Birth; Group Prenatal Care; Respectful Care; Patient Satisfaction; Prenatal Depression and Anxiety; Low Income; Health Inequity; Prenatal Care; Person-Centered Care
MeSH Terms: conditions — Premature Birth; Depression; Anxiety Disorders; Depression, Postpartum; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glow! Group Prenatal Care (Active Comparator): Group prenatal care with wrap around services.
  Interventions: Other: Glow! Group Prenatal Care
- Individual Prenatal Care- CPSP (Active Comparator): Individual prenatal care with supplemental services covered by CPSP.
  Interventions: Other: Individual Prenatal Care with CPSP

INTERVENTIONS:
Other: Glow! Group Prenatal Care — Glow! is an enhanced group prenatal care model that offers co-located social services provided by established community programs with independent funding streams targeting low-income families. The Glow! group prenatal care model pairs a trained facilitator with a licensed prenatal care practitioner from a practice site to provide billable prenatal care to the practice's own patients. Over the course of 8-10 sessions, 10-12 women (within a 6- week gestational age range) receive prenatal medical care, risk assessments, and social support, and gain knowledge and skills related to pregnancy, birth, and parenting.
  Arms: Glow! Group Prenatal Care
Other: Individual Prenatal Care with CPSP — Comprehensive Perinatal Services Program (CPSP) is a state-funded program for Medi-Cal eligible families to receive enhanced care and service coordination. Participants assigned to CPSP individual care may participate in the CPSP assessments with a Comprehensive Perinatal Health Worker at their prenatal care site, where individual prenatal care will be provided
  Arms: Individual Prenatal Care- CPSP

SUMMARY:
This is a randomized comparative effectiveness study of two forms of enhanced prenatal care among 657 Medi-Cal eligible pregnant individuals in Fresno, California. The goal is to see whether group prenatal care with wrap around services versus individual prenatal care supplemented by services covered by the California Department of Public Health Comprehensive Perinatal Services Program (CPSP) results in less depression and anxiety, and more respectful, more person-centered maternity care and lower rates of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 24 weeks gestation at enrollment
* Eligible for Medi-Cal (at or below 213% of the federal poverty level)
* Speak English or Spanish

Exclusion Criteria:

* Unavailable to attend group prenatal care sessions
* Not planning to continue prenatal care with site provider
* Cannot legally consent to participate in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in Patient Health Questionnaire (PHQ-9) Score | Collected from study enrollment to three months postpartum
  Changes in depressive symptom severity from baseline to postpartum. Assessed using the Patient Health Questionnaire (PHQ-9), administered in-person at baseline and during telephone interview at three months postpartum. Total score ranges from 0-27 with higher scores indicating more severe depression.
Person-centered prenatal care | Collected during third trimester
  This outcome focuses on the extent to which the participants feels their prenatal care was person centered.
  The title of the measure is Person Centered Prenatal Care (primary). This measurement tool is a questionnaire that includes series of items that were developed in collaboration with community members to measure their experience of care. In addition to the overall score, the scale includes three subscales identified as important by community members: dignity and respect, communication and autonomy, and responsive and supportive care. The measures have been validated in several languages.
  The total scores range from 0-100 with higher scores indicating the receipt of more person centered care.
Preterm birth | 0-12 weeks after delivery
  Whether the participant had a baby born less than 37 weeks gestation, as noted in the participant's medical record.

SECONDARY OUTCOMES:
Changes in anxiety symptom severity | Collected from study enrollment to three months postpartum
  Changes in anxiety symptom severity from baseline to postpartum. Assessed using the 7-item Generalized Anxiety Disorder (GAD-7) scale, administered in-person at baseline and during telephone interview at three months postpartum.
  The total scores range from 0-21 with higher scores indicating more severe anxiety.
Perceptions of respectful/disrespectful maternity care | Collected at three months postpartum
  Extent to which the participant feels that the maternity care they received was respectful. Assessed using the Mothers on Respect Index (MORi), administered during telephone interview or in-person at third trimester and three months postpartum.
  The total scores range from 14-84 with higher scores indicating a higher level of respect.
Satisfaction with prenatal care | Collected during third trimester and at three months postpartum
  Extent to which the participant feels satisfied with the prenatal care they received. Assessed using the Prenatal Care Satisfaction Scale, administered during telephone interview or in-person interview at third trimester and three months postpartum.
  The total scores range from 0-100 with higher scores indicating higher levels of satisfaction.
Gestational age at delivery | 0-12 weeks after delivery
  The gestation age at which the baby was born (number of weeks), as noted in the participant's medical record.
Person Centered Maternity Care as measured at 3 months postpartum. | 3 months postpartum
  Extent to which birthing person feels their prenatal and birthing experience was person centered, as measured by the Person-Centered Maternity Care scale.
  This measure focuses on the extent to which the participants feels their prenatal and maternity/birthing care was person centered.
  The title of the measure is Person Centered Maternity Care. This measurement tool is a questionnaire that includes series of items that were developed in collaboration with community members to measure their experience of care. In addition to the overall score, the scale includes three subscales identified as important by community members: dignity and respect, communication and autonomy, and responsive and supportive care. The measures have been validated in several languages.
  The total scores range from 0-100 with higher scores indicating the receipt of more person centered care.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kuppermann, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Central Valley Health Policy Institute, Fresno, California
  - UCSF, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Raube K, Handler A, Rosenberg D. Measuring satisfaction among low-income women: a prenatal care questionnaire. Matern Child Health J. 1998 Mar;2(1):25-33. doi: 10.1023/a:1021841508698. PMID 10728256
- [Background] Vedam S, Stoll K, Rubashkin N, Martin K, Miller-Vedam Z, Hayes-Klein H, Jolicoeur G; CCinBC Steering Council. The Mothers on Respect (MOR) index: measuring quality, safety, and human rights in childbirth. SSM Popul Health. 2017 Jan 19;3:201-210. doi: 10.1016/j.ssmph.2017.01.005. eCollection 2017 Dec. PMID 29349217
- [Background] Peek ME, Nunez-Smith M, Drum M, Lewis TT. Adapting the everyday discrimination scale to medical settings: reliability and validity testing in a sample of African American patients. Ethn Dis. 2011 Autumn;21(4):502-9. PMID 22428358
- [Background] Krieger N, Smith K, Naishadham D, Hartman C, Barbeau EM. Experiences of discrimination: validity and reliability of a self-report measure for population health research on racism and health. Soc Sci Med. 2005 Oct;61(7):1576-96. doi: 10.1016/j.socscimed.2005.03.006. Epub 2005 Apr 21. PMID 16005789
- [Derived] Kuppermann M, Pressman A, Coleman-Phox K, Afulani P, Blebu B, Carraway K, Butcher BC, Curry V, Downer C, Edwards B, Felder JN, Fontenot J, Garza MA, Karasek D, Lessard L, Martinez E, McCulloch CE, Oberholzer C, Ramirez GR, Tesfalul M, Wiemann A. A randomized comparative-effectiveness study of two enhanced prenatal care models for low-income pregnant people: Engaging Mothers & Babies; Reimagining Antenatal Care for Everyone (EMBRACE). Contemp Clin Trials. 2024 Aug;143:107568. doi: 10.1016/j.cct.2024.107568. Epub 2024 May 14. PMID 38750950
- [Derived] Felder JN, Afulani PA, Coleman-Phox K, Omowale SS, McCulloch CE, Lessard L, Kuppermann M. Pregnancy-related COVID worry, depressive symptom severity, and mediation through sleep disturbance in a low-income, primarily Latinx population in California's Central valley. J Psychiatr Res. 2023 Jan;157:96-103. doi: 10.1016/j.jpsychires.2022.11.019. Epub 2022 Nov 23. PMID 36459760